CLINICAL TRIAL: NCT03003390
Title: Prevention of Central Venous Catheter-associated Thrombosis in Critically Ill Children: A Multicenter Phase 2b Trial
Brief Title: Catheter-Related Early Thromboprophylaxis With Enoxaparin (CRETE) Trial
Acronym: CRETE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Met protocol defined stopping rule for futility
Sponsor: Yale University (Other)
Collaborators: St. Louis Children's Hospital (Other); Dell Children's Medical Center of Central Texas (Other); Children's Hospital and Health System Foundation, Wisconsin (Other); Weill Medical College of Cornell University (Other); Maria Fareri Children's Hospital (Unknown); University of Rochester (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1302011506; 1R21HD089131-01A1 (NIH)
Record Dates: First submitted 2016-12-19; First posted 2016-12-28 (Estimated); Results first posted 2020-07-13 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-03

CONDITIONS: Deep Venous Thrombosis
Keywords: child; critical illness; venous thromboembolism; enoxaparin; thrombin generation
MeSH Terms: conditions — Venous Thrombosis; Critical Illness; Venous Thromboembolism | interventions — Enoxaparin

STUDY DESIGN:
Intervention Model Description: Eligible subjects will be randomized 1:1 to treatment or control.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Prophylaxis with enoxaparin (Experimental): A clinical nurse will administer enoxaparin subcutaneously <24 hours after insertion of the central venous catheter and then give enoxaparin subcutaneously every 12 hours until the removal of the catheter.
  Interventions: Drug: Enoxaparin
- Control arm (No Intervention): Participants randomized to the control arm will receive no 'placebo' intervention.

INTERVENTIONS:
Drug: Enoxaparin — The clinical nurse will give enoxaparin subcutaneously every 12 hours at the currently used starting dose of 0.75 mg/kg for children ≤2 months old or 0.5 mg/kg (maximum of 40 mg) for older children. The 1st dose will be given <24 hours after insertion of the catheter. Doses will be adjusted to target an anti-Xa level of 0.2-0.5 IU/mL.
  Other Names: Lovenox
  Arms: Prophylaxis with enoxaparin

SUMMARY:
The purpose of this phase 2a, multi-center, randomized controlled study, is to explore the efficacy of early prophylaxis against catheter-associated deep venous thrombosis (CADVT) in critically ill children.

DETAILED DESCRIPTION:
Critical illness and the presence of a central venous catheter (CVC) are the most important risk factors for deep venous thrombosis (DVT) in children. Catheter-associated thrombosis (CADVT) is highly prevalent and associated with poor outcomes in critically ill children. Yet, based on underpowered pediatric trials, prophylaxis against CADVT is not recommended in children. The recommendation to provide prophylaxis against thrombosis in critically ill adults should not be applied to children because the hemostatic system and co-morbidities vastly differ between age groups. Pivotal trials are urgently needed to determine whether prophylaxis can prevent CADVT and its complications in critically ill children. However, the timing and extent of reduction in thrombin generation, the biochemical goal of prophylaxis, needed to prevent CADVT in children are unclear. The goal of this application is to explore the efficacy of early prophylaxis against CADVT in critically ill children. Aim 1 is to obtain preliminary evidence on the effect of early prophylaxis on the incidence of CADVT in critically ill children. Based on the natural history of CADVT, we hypothesize that among critically ill children, prophylaxis administered <24 hours after catheter insertion decreases the incidence of ultrasound-diagnosed CADVT compared with no prophylaxis. In this phase 2a trial, children admitted to the intensive care unit with a newly inserted central venous catheter will receive enoxaparin adjusted according to anti-Xa activity, a control group will not receive enoxaparin adjusted according to anti-Xa activity. Enoxaparin has become the "standard" pediatric anticoagulant for prophylaxis despite the absence of conclusive data. We will use Bayesian approach to determine whether further trials are warranted. Aim 2 is to evaluate the effect of an anti-Xa activity-directed prophylactic strategy on thrombin generation in critically ill children. We hypothesize that among critically ill children, standard prophylactic dose of enoxaparin adjusted by anti-Xa activity reduces thrombin generation to <700 nanomolar-minute (nM.min), as measured by endogenous thrombin potential (ETP). In non-critically ill adults, prophylactic dose of enoxaparin proven to prevent DVT reduces ETP to <700 nM.min. Endogenous thrombin potential is the best available measure of thrombin generation. We will measure endogenous thrombin potential and anti-Xa activity at multiple time points then examine their relationship in all children enrolled in the phase 2a trial. The proposed research challenges the current paradigm on prophylaxis against CADVT in children. High quality evidence is needed to prevent CADVT and its complications in this vulnerable population.

ELIGIBILITY:
Inclusion Criteria

1. Untunneled CVC inserted in the internal jugular or femoral vein within the past 24 hours
2. Child anticipated to stay in the pediatric intensive care unit ≥48 hours
3. CVC anticipated to be required for ≥24 hours
4. >36 weeks corrected gestational age to <18 years old

Exclusion Criteria

1. Coagulopathy (i.e., international normalized ratio >2.0, activated partial thromboplastin time >50 seconds or platelet count <50,000/mm3)
2. Known bleeding disorder
3. Clinically relevant bleeding as defined by the International Society on Thrombosis and Hemostasis (i.e., Hb decreased ≥2 g/dl in 24 hours, required medical or surgical intervention to restore hemostasis, or in a critical organ system [i.e., retroperitoneum, pulmonary, intracranial or central nervous system])
4. <60 days from a clinically relevant bleeding as defined above
5. <7 days after trauma or surgery
6. Anticipated surgery within 48 hours after insertion of the CVC
7. Renal failure (i.e., creatinine clearance <30 mL/min)
8. Presence of epidural catheter
9. Currently taking an antithrombotic agent (e.g., low molecular weight heparin (LMWH), unfractionated heparin (UFH) at therapeutic doses, Coumadin or aspirin)
10. Radiologically documented DVT at the site of insertion of the CVC in the previous 6 weeks
11. Known hypersensitivity to heparin or its components, including pork products
12. History of heparin-induced thrombocytopenia (HIT) (i.e., positive serotonin release assay)
13. Currently pregnant
14. Currently lactating
15. Prior enrollment in the study
16. Limitation of care

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2017-04-05 (Actual); Primary Completion 2019-08-16 (Actual); Study Completion 2019-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: E. Vincent S Faustino, MD, MHS, Principal Investigator — Associate Professor of Pediatrics, Yale School of Medicine
Locations (6):
- United States (6):
  - Yale University Yale New Haven Health, New Haven, Connecticut
  - Saint Louis Children's Hospital-Washington University School of Medicine-, St Louis, Missouri
  - Weill Cornell Medicine, New York, New York
  - University of Rochester Medical Center-Golisano Children's Hospital-, Rochester, New York
  - Maria Fareri Children's Hospital, Valhalla, New York
  - Children's Hospital of Wisconsin/Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Faustino EVS, Raffini LJ, Hanson SJ, Cholette JM, Pinto MG, Li S, Kandil SB, Nellis ME, Shabanova V, Silva CT, Tala JA, McPartland T, Spinella PC; for the CRETE Trial Investigators and the Pediatric Critical Care Blood Research Network (BloodNet) of the Pediatric Acute Lung Injury and Sepsis Investigators Network (PALISI); CRETE Trial Investigators: Clinical Coordinating Center:; and; Data Coordinating Center:; and; Outcomes Adjudication Committee:; and; Data and Safety Monitoring Board:; and; Independent Safety Monitor:; and; Children's Hospital Wisconsin:; and; Dell Children's Medical Center:; and; Maria Fareri Children's Hospital:; and; St. Louis Children's Hospital:; and; University of Rochester Golisano Children's Hospital:; and; Weill Cornell Medical Center:; and; and Yale-New Haven Children's Hospital:; and; for the CRETE Trial Investigators and the Pediatric Critical Care Blood Research Network (BloodNet) of the Pediatric Acute Lung Injury and Sepsis Investigators Network (PALISI) and CRETE Trial Investigators: Clinical Coordinating Center: and and and Data Coordinating Center: and and and Outcomes Adjudication Committee: and and and Data and Safety Monitoring Board: and and and Independent Safety Monitor: and and and Children's Hospital Wisconsin: and and and Dell Children's Medical Center: and and and Maria Fareri Children's Hospital: and and and St. Louis Children's Hospital: and and and University of Rochester Golisano Children's Hospital: and and and Weill Cornell Medical Center: and and and and Yale-New Haven Children's Hospital: and and. Age-Dependent Heterogeneity in the Efficacy of Prophylaxis With Enoxaparin Against Catheter-Associated Thrombosis in Critically Ill Children: A Post Hoc Analysis of a Bayesian Phase 2b Randomized Clinical Trial. Crit Care Med. 2021 Apr 1;49(4):e369-e380. doi: 10.1097/CCM.0000000000004848. PMID 33566465
- [Derived] Faustino EVS, Shabanova V, Raffini LJ, Kandil SB, Li S, Pinto MG, Cholette JM, Hanson SJ, Nellis ME, Silva CT, Chima R, Sharathkumar A, Thomas KA, McPartland T, Tala JA, Spinella PC; CRETE Trial Investigators and the Pediatric Critical Care Blood Research Network (BloodNet) of the Pediatric Acute Lung Injury and Sepsis Investigators Network (PALISI). Efficacy of Early Prophylaxis Against Catheter-Associated Thrombosis in Critically Ill Children: A Bayesian Phase 2b Randomized Clinical Trial. Crit Care Med. 2021 Mar 1;49(3):e235-e246. doi: 10.1097/CCM.0000000000004784. PMID 33372745

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One participant in the enoxaparin group was enrolled during a single arm phase and not included in the analysis.
Period: Overall Study
Arm/Group | Prophylaxis With Enoxaparin | Control Arm
Started | 27 | 24
Completed | 23 | 24
Not Completed | 4 | 0
Not completed — Physician Decision | 2 | 0
Not completed — Parent refused intervention | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prophylaxis With Enoxaparin | Control Arm | Total
Number analyzed (Participants) | 27 | 24 | 51
Age, Customized [Count of Participants; unit: Participants]
  <1 year old | 12 | 12 | 24
  1-13 years old | 13 | 10 | 23
  >13 years old | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 12 | 28
  Male | 11 | 12 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 10
  Not Hispanic or Latino | 22 | 19 | 41
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 7 | 13
  White | 20 | 17 | 37
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Size of Central Venous Catheter (CVC) [Count of Participants; unit: Participants] — The size of the CVC may affect the risk of CVC-associated DVT. Larger diameter of the CVC, i.e. higher F, particular relative to the size of the central vein has been associated with higher risk of DVT. The size of the CVC was determined by the clinical team.
  Participants
    3 French (F) | 0 | 2 | 2
    4 F | 13 | 11 | 24
    5 F | 10 | 10 | 20
    7 F | 4 | 1 | 5
Number of Lumens of CVC [Count of Participants; unit: Participants]
  1 | 0 | 2 | 2
  2 | 15 | 12 | 27
  3 | 12 | 10 | 22
Site of Insertion of CVC [Count of Participants; unit: Participants]
  Left Femoral | 4 | 4 | 8
  Right Internal Jugular | 15 | 13 | 28
  Right Femoral | 8 | 7 | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Central Venous Catheter (CVC)- Associated Deep Vein Thrombosis (DVT)
Description: Thrombus in the central vein where the CVC was inserted that is clinically suspected then confirmed radiologically, an incidental radiologic finding, or diagnosed with the study-related active surveillance ultrasound
Time Frame: Up to removal of CVC, an average of 6 days
Measure: Count of Participants; unit: Participants
Arm/Group | Prophylaxis With Enoxaparin | Control Arm
Number analyzed (Participants) | 23 | 24
Participants | 7 | 13
Statistical Analysis 1: Comparison: Prophylaxis With Enoxaparin vs Control Arm; Test type: Superiority; Posterior probabilities = 0.09; Using informative priors of B(1, 1) on the enoxaparin arm and B(18, 82) on the usual care arm, the risks of CADVT were 0.32 (95% CrI: 0.16, 0.51) in the enoxaparin arm and 0.25 (95% CrI: 0.18, 0.33) in the usual care arm. The posterior probability that the absolute difference in the risk of CADVT was lower by 0.06 in the enoxaparin arm was 9.1%. Using minimally informative priors, the risk ratio of CADVT with enoxaparin was 0.55 (95% CrI: 0.24, 1.11)

2. Primary Outcome: Endogenous Thrombin Potential
Description: An established measure of coagulation status and is the best method to measure thrombin generation. It directly measures the amount of thrombin generation over time capturing the effects of natural (i.e., subject's coagulation status) and pharmacological (e.g., enoxaparin) pro- and anticoagulants. Endogenous thrombin potential is measured using thrombin generation assay.
Time Frame: Day of, day after and day 4 after insertion of the CVC
Population: The numbers analyzed on the day after CVC insertion and four days after CVC insertion differ from the overall number of participants. Participants were excluded if the CVC was removed or if blood was not drawn.
Measure: Median (Inter-Quartile Range); unit: Nanomolar-minute (nM.min)
Arm/Group | Prophylaxis With Enoxaparin | Control Arm
Number analyzed (Participants) | 27 | 24
Nanomolar-minute (nM.min)
  Day of CVC Insertion | 919.7 [418.71 to 1150.77] | 1035.6 [800.22 to 1455.05]
  Day After CVC Insertion: number analyzed (Participants) | 24 | 22
  Day After CVC Insertion | 851.19 [627.31 to 995.98] | 896.58 [433.9 to 1331.03]
  Day 4 After CVC Insertion: number analyzed (Participants) | 20 | 20
  Day 4 After CVC Insertion | 826.97 [0 to 1131.7] | 969.89 [605.35 to 1302.95]
Statistical Analysis 1: Comparison: Prophylaxis With Enoxaparin vs Control Arm; Test type: Superiority; p = 0.22, Linear mixed effects model

3. Secondary Outcome: Number With Other Thromboembolic Events
Description: Thrombus in the deep vein of any extremity or PE that is clinically suspected then confirmed radiologically, an incidental radiologic finding, excluding DVT diagnosed with the study-related active surveillance ultrasound
Time Frame: Up to removal of CVC, an average of 6 days
Measure: Count of Participants; unit: Participants
Arm/Group | Prophylaxis With Enoxaparin | Control Arm
Number analyzed (Participants) | 27 | 24
Participants | 1 | 1
Statistical Analysis 1: Comparison: Prophylaxis With Enoxaparin vs Control Arm; Test type: Superiority; p = 1.00, Fisher Exact

4. Secondary Outcome: Length of Stay in the Pediatric Intensive Care Unit in Days
Description: Duration of stay in the pediatric intensive care unit from the day of enrollment
Time Frame: Up to day of discharge from the pediatric intensive care unit, an average of 10 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Prophylaxis With Enoxaparin | Control Arm
Number analyzed (Participants) | 27 | 24
days | 12 [6 to 22] | 8 [4 to 16]
Statistical Analysis 1: Comparison: Prophylaxis With Enoxaparin vs Control Arm; Test type: Superiority; p = 0.31, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Length of Stay in the Hospital
Description: Duration of stay in the hospital from the day of enrollment
Time Frame: Up to day of discharge from the hospital, an average of 18 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Prophylaxis With Enoxaparin | Control Arm
Number analyzed (Participants) | 27 | 24
days | 16 [6 to 35] | 16 [7 to 23]
Statistical Analysis 1: Comparison: Prophylaxis With Enoxaparin vs Control Arm; Test type: Superiority; p = 0.58, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Number With Clinically Relevant Bleeding
Description: Bleeding that is fatal, associated with a decrease in hemoglobin by ≥2 g/dl in 24 hours, requires medical or surgical intervention to restore hemostasis, or is in the retroperitoneum, pulmonary, intracranial or central nervous system as defined by International Society of Thrombosis and Haemostasis
Time Frame: Up to 30 hours after the last enoxaparin dose
Measure: Count of Participants; unit: Participants
Arm/Group | Prophylaxis With Enoxaparin | Control Arm
Number analyzed (Participants) | 27 | 24
Participants | 1 | 0
Statistical Analysis 1: Comparison: Prophylaxis With Enoxaparin vs Control Arm; Test type: Superiority; p = 1.00, Fisher Exact

7. Secondary Outcome: Number With Laboratory Confirmed Heparin-induced Thrombocytopenia
Description: Heparin-induced thrombocytopenia that is diagnosed with a positive serotonin release assay
Time Frame: Up to removal of CVC, an average of 6 days
Population: None of the participants experienced this outcome; hence, a statistical analysis was not performed.
Measure: Count of Participants; unit: Participants
Arm/Group | Prophylaxis With Enoxaparin | Control Arm
Number analyzed (Participants) | 27 | 24
Participants | 0 | 0

8. Secondary Outcome: Number of Mortality
Description: In-hospital mortality during the subject's admission
Time Frame: Up to day of discharge from the hospital, average of 18 days
Measure: Count of Participants; unit: Participants
Arm/Group | Prophylaxis With Enoxaparin | Control Arm
Number analyzed (Participants) | 27 | 24
Participants | 5 | 2
Statistical Analysis 1: Comparison: Prophylaxis With Enoxaparin vs Control Arm; Test type: Superiority; p = 0.43, Fisher Exact

9. Secondary Outcome: Number of Enrolled Eligible Children
Description: Number of eligible children enrolled in the study.
Time Frame: Up to 24 hours after insertion of CVC
Measure: Count of Participants; unit: Participants
Groups:
- Eligible Children: Children eligible to participate in this study.
Arm/Group | Eligible Children
Number analyzed (Participants) | 164
Participants | 51

10. Secondary Outcome: Time to 1st Dose of Enoxaparin
Description: Time to first dose of enoxaparin
Time Frame: Up to 48 hours after insertion of CVC
Measure: Median (Inter-Quartile Range); unit: hours from insertion of CVC
Groups:
- Prophylaxis With Enoxaparin: Participants in the treatment arm received enoxaparin.
Arm/Group | Prophylaxis With Enoxaparin
Number analyzed (Participants) | 27
hours from insertion of CVC | 21.1 [14.7 to 23.5]

11. Secondary Outcome: Time to Target Anti-Xa Activity
Description: Time from insertion of the CVC to time that anti-Xa activity was within 0.2-0.5 IU/mL.
Time Frame: Up to removal of CVC, an average of 6 days
Population: This outcome measure is only applicable to subjects in the enoxaparin arm because the control arm did not receive enoxaparin for which anti-Xa activity is used to titrate the dose. Only 12 participants in the enoxaparin arm achieved the target anti-Xa activity.
Measure: Median (Inter-Quartile Range); unit: hours from insertion of CVC
Groups:
- Prophylaxis With Enoxaparin: Children were treated with enoxaparin
Arm/Group | Prophylaxis With Enoxaparin
Number analyzed (Participants) | 12
hours from insertion of CVC | 70.4 [47.4 to 92.2]

12. Secondary Outcome: Number of Missed Doses of Enoxaparin
Description: Number of doses of enoxaparin that were not administered. This outcome measure was only applicable to the enoxaparin arm.
Time Frame: Up to removal of CVC, an average of 6 days
Measure: Number; unit: Doses of enoxaparin
Units Other Than Participants: Doses
Arm/Group | Prophylaxis With Enoxaparin
Number analyzed (Participants) | 27
Number analyzed (Doses) | 272
Doses of enoxaparin | 8

13. Secondary Outcome: Number of Children With Ultrasound
Description: Number of children in whom ultrasound was not performed.
Time Frame: Up to 24 hours after removal of CVC
Measure: Count of Participants; unit: Participants
Groups:
- All Enrolled Children: All children who participated in the study
Arm/Group | All Enrolled Children
Number analyzed (Participants) | 51
Participants | 47

ADVERSE EVENTS:
Time Frame: From hospital admission to day of discharge for death, up to 60 days.
Arm/Group | Prophylaxis With Enoxaparin | Control Arm
All-Cause Mortality (participants affected / at risk) | 5/27 | 2/24
Serious Adverse Events (participants affected / at risk) | 2/27 | 0/24
Other Adverse Events (participants affected / at risk) | 9/27 | 6/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prophylaxis With Enoxaparin (N=27) | Control Arm (N=24)
acute kidney injury (Renal and urinary disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Prophylaxis With Enoxaparin (N=27) | Control Arm (N=24)
Acidosis (Metabolism and nutrition disorders) | 3 | 1
Anemia (Blood and lymphatic system disorders) | 5 | 3
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Edema trunk (General disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
General disorders and administration site conditions - Other, specify (General disorders) | 0 | 1
Hematuria (Renal and urinary disorders) | 1 | 1
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Oral hemorrhage (Gastrointestinal disorders) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 1 | 0
Tracheitis (Infections and infestations) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2017-08-25): https://cdn.clinicaltrials.gov/large-docs/90/NCT03003390/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2017-08-22): https://cdn.clinicaltrials.gov/large-docs/90/NCT03003390/Prot_SAP_001.pdf